CLINICAL TRIAL: NCT00198445
Title: Efficacy and Safety of Topical Bromfenac Ophthalmic Solution, 0.1% vs. Placebo for Treatment of Ocular Inflammation Following Cataract Surgery
Brief Title: Safety and Efficacy Study of Topical Bromfenac Versus Placebo to Treat Ocular Inflammation After Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISTA-BR-CS001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Postoperative Complications; Cataract
Keywords: Cataract Extraction; Anti-Inflammatory Agents, Non-Steroidal
MeSH Terms: conditions — Postoperative Complications; Cataract | interventions — bromfenac

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bromfenac (Experimental): Topical bromfenac ophthalmic solution 0.1%
  Interventions: Drug: Bromfenac
- Placebo (Placebo Comparator): Vehicle of bromfenac
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bromfenac — One drop in study eye every 12 hours for 14 days
  Arms: Bromfenac
Drug: Placebo — One drop in study eye every 12 hours for 14 days
  Arms: Placebo

SUMMARY:
The primary objective of this study was to investigate the efficacy of bromfenac sodium ophthalmic solution 0.09% for treatment of post-operative ocular inflammation in subjects who undergo cataract extraction and intraocular lens implantation. The secondary objective was to investigate the safety and tolerability of the same.

ELIGIBILITY:
Inclusion Criteria:

* Cataract surgery
* Summed ocular inflammation score (anterior chamber cell score plus flare score) of >/= 3, 24 hours after the cataract extraction
* Agreed to avoid disallowed medications (meds) throughout the duration of the study

Exclusion Criteria:

* Use of or need for non-steroidal anti-inflammatory agents (NSAIDs), steroids, anticoagulants, or other specific meds prohibited by the protocol
* Uncontrolled chronic ocular or systemic disease, active corneal pathology or scarring noted in either eye (except keratopathy, allowed in non-study eye)
* Extraocular/intraocular inflammation in either eye
* Clinically significant (WHO CTC Grade 1 or greater) liver function tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2003-05; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Ocular Inflammation Score | Visit 4 (Day 15)
  Cleared ocular inflammation in the study eye, defined as summed ocular inflammation score (SOIS) of 1 or less (anterior chamber cell score plus flare score, each measured on a 5-point scale) 0=none

SECONDARY OUTCOMES:
Mean Ocular Inflammation Score | At each Visit 2 (Day3), Visit 3 (Day 8), Visit 4 (Day 15), Visit 5 (Day 22)
  Mean change from baseline in SOIS at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Grillone, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (39):
- United States (39):
  - Harold A Helms, MD, Birmingham, Alabama
  - Eye Care Arkansas, PA, Little Rock, Arkansas
  - UCI, Department of Ophthalmology, Irvine, California
  - Anesthetic Eye Care Institute, Newport Beach, California
  - Richard A Lewis, MD, Sacramento, California
  - Eye Care of San Diego, San Diego, California
  - Santa Clara Valley Medical Center, San Jose, California
  - E Randy Craven, MD, Littleton, Colorado
  - The Eye Care Group, New Haven, Connecticut
  - Cohen Laser Vision Center, Boca Raton, Florida
  - Brandon Cataract Center & Eye Clinic, Brandon, Florida
  - Marvin E Greenberg, MD, PA, Tamarac, Florida
  - Jack Daubert, MD, West Palm Beach, Florida
  - Advanced Eye Care, PC, Fort Oglethorpe, Georgia
  - Saltzer Medical Group, PA, Nampa, Idaho
  - Donald E Beahm, MD, Great Bend, Kansas
  - Cincinnati Eye Institute NKY, Edgewood, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Stevenson Medical Surgical Eye Center, New Orleans, Louisiana
  - Cornea Consultants, Boston, Massachusetts
  - Great Lakes Eye Care, Saint Joseph, Michigan
  - Hunkeler Eye Institute, Kansas City, Missouri
  - Arthur J Weinstein, MD, Albuquerque, New Mexico
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Horizon Eye Care, Charlotte, North Carolina
  - Dean A McGee Eye Institute, Oklahoma City, Oklahoma
  - The Eye Institute, Tulsa, Oklahoma
  - Casey Eye Institute, Portland, Oregon
  - Eye Health Northwest, Portland, Oregon
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Middle Tennessee Eye Associates, Cookeville, Tennessee
  - Texan Eye Care PA, Austin, Texas
  - Ophthalmology Service, Brooke Army Medical Center, Fort Sam Houston, Texas
  - Ophthalmology Visual Science, Galveston, Texas
  - Houston Eye Associates, Houston, Texas
  - David G Shulman, MD, San Antonio, Texas
  - Central Texas Eye Center, San Marcos, Texas
  - Virginia Eye Consultants, Norfolk, Virginia